CLINICAL TRIAL: NCT01783093
Title: An Evaluation of Tricuspid Regurgitant Jet Velocity as an Independent Marker for Mortality in Patients With Sickle Cell Anemia: A Retrospective Data Review
Brief Title: Tricuspid Regurgitant Jet Velocity as an Independent Marker for Mortality in Sickle Cell Anemia
Status: Completed | Type: Observational
Sponsor: Namita Sood (Other)
Responsible Party: Sponsor-Investigator, Namita Sood, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Other Study IDs: 2009H0269
Record Dates: First submitted 2011-08-17; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Sickle Cell Anemia; Pulmonary Hypertension
MeSH Terms: conditions — Anemia, Sickle Cell; Hypertension, Pulmonary | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Sickle cell and pulmonary hypertension
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Collection of data from existing medical records

SUMMARY:
The purpose of this study is to evaluate patients with pulmonary hypertension and sickle cell disease who have had multiple echocardiograms. Previous studies have shown that an elevated tricuspid jet (TR) regurgitant velocity on echo in this population is a predictor of mortality. This initial data only examined an isolated TR jet velocity. It was presumed that the mortality was related to pulmonary hypertension.

It is the aim of this study to retrospectively evaluate patients who have had multiple echocardiograms and to determine if patients who had either a normalization of their TR jet velocity on a subsequent echo or had no evidence of pulmonary hypertension on right heart catheterization had a similar mortality rate to those with persistently elevated TR jet velocity.

ELIGIBILITY:
To limit bias in this study all patients that with sickle cell anemia and pulmonary hypertension with the pre-specified data required will be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients records will be extracted from the complete medical record at OSUMC
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
A retrospective review on patients who have had multiple echocardiograms to determine if patients with a normalization of TR Jet Velocity have changes in risk of death compared with those who do not have normalization of TR Jet Velocity. | Up to 20 years
  Any subject's who meet criteria and have multiple echocardiograms may be included.

CONTACTS AND LOCATIONS:
Overall Officials: Namita Sood, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- [Background] Gladwin MT, Sachdev V, Jison ML, Shizukuda Y, Plehn JF, Minter K, Brown B, Coles WA, Nichols JS, Ernst I, Hunter LA, Blackwelder WC, Schechter AN, Rodgers GP, Castro O, Ognibene FP. Pulmonary hypertension as a risk factor for death in patients with sickle cell disease. N Engl J Med. 2004 Feb 26;350(9):886-95. doi: 10.1056/NEJMoa035477. PMID 14985486
- [Background] Gladwin MT, Vichinsky E. Pulmonary complications of sickle cell disease. N Engl J Med. 2008 Nov 20;359(21):2254-65. doi: 10.1056/NEJMra0804411. No abstract available. PMID 19020327
- [Background] Ballas SK. The cost of health care for patients with sickle cell disease. Am J Hematol. 2009 Jun;84(6):320-2. doi: 10.1002/ajh.21443. No abstract available. PMID 19415728
- [Background] Farber HW, Loscalzo J. Pulmonary arterial hypertension. N Engl J Med. 2004 Oct 14;351(16):1655-65. doi: 10.1056/NEJMra035488. No abstract available. PMID 15483284
- [Background] De Castro LM, Jonassaint JC, Graham FL, Ashley-Koch A, Telen MJ. Pulmonary hypertension associated with sickle cell disease: clinical and laboratory endpoints and disease outcomes. Am J Hematol. 2008 Jan;83(1):19-25. doi: 10.1002/ajh.21058. PMID 17724699